CLINICAL TRIAL: NCT05302401
Title: Effect of Intrapartum Continuous Midwife Support on Maternal and Neonatal Stress Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: M_aslan
Record Dates: First submitted 2022-01-30; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-01

CONDITIONS: Labor Complication; Midwife; Stress; Labor Pain
Keywords: Continuous midwife support; Midwife; Labour support; Stress; Neonatal; Intrapartum; Cortisol; Saliva
MeSH Terms: conditions — Obstetric Labor Complications; Labor Pain | interventions — Prenatal Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women receiving uninterrupted midwife support during the intrapartum period (Experimental): 28. - Visual Analog Scale will be applied to determine the Wijma Birth Expectation/Experience (W-DEQ A) Scale and birth fear in order to determine the birth fears of pregnant women in the 36th week. During outpatient checks, the first saliva cortisol samples will be taken by researcher Meserret Aslan between 8:30 and 09:00 in the morning. Researcher Meserret Aslan will provide six hours of online pregnancy training to pregnant women in the experimental group and provide uninterrupted midwife support during the intrapartum period.Within the first half hour of postpartum after birth, saliva cortisol samples of women will be repeated by researcher Meserret Aslan. Between the 24th and 72nd hours before postpartum discharge procedures take place, saliva cortisol samples of women will be taken for the last time by researcher Meserret Aslan from the experimental group.
  Interventions: Behavioral: intrapartum uninterrupted midwife support
- Women who do not receive uninterrupted midwife support during the intrapartum period (No Intervention): Between the 28th and 36th weeks, the pregnancy diagnosis form will be applied by the researcher to the pregnant women in the control group. 28. - Visual Analog Scale will be applied to determine the Wijma Birth Expectation/Experience (W-DEQ A) Scale and birth fear in order to determine the birth fears of pregnant women in the 36th week. During outpatient checks, the first saliva cortisol samples will be taken by researcher Meserret Aslan between 8:30 and 09:00 in the morning. After birth, postpartum from control groups will be repeated by researcher Meserret Aslan in the first half hour. Between the 24th and 72nd hours before postpartum discharge procedures take place, saliva cortisol samples of women will be taken for the last time by researcher Meserret Aslan from the control groups.

INTERVENTIONS:
Behavioral: intrapartum uninterrupted midwife support — Prenatal women will be trained about the birth process and psychological and physical support will be provided to women during childbirth. Among these supports, healthy women will be exercised during the labor action, given positions that facilitate childbirth, their hands will be held when they need them, their oral intake will not be restricted, and warm showers will be applied according to their wishes. (These applications can be increased.)
  Other Names: Prenatal education
  Arms: Women receiving uninterrupted midwife support during the intrapartum period

SUMMARY:
This study aims to provide strong A-level evidence to the literature by supporting the maternal and fetal results of continuous midwife support together with saliva cortisol level measurements. As a result of this study, it is expected that women who receive intrapartum continuous midwife support and their babies have lower saliva cortisol levels than women in the control group, women who receive intrapartum continuous midwife support experience less fear, and women who receive intrapartum uninterrupted midwife support are expected to have lower intervention rates in their births. If the existing hypotheses are accepted, it is aimed to expand the practice of intrapartum continuous midwife support. Although pregnancy, childbirth and postpartum period are a physiological process, it is an important source of stress brought on by physical and hormonal changes for women's life. Uninterrupted midwife support in women who will give birth is associated with more vaginal births and fewer negative birth experiences. Uninterrupted midwife care also has higher female satisfaction, less intervention and lower maintenance costs. Therefore, evidence-based practices are needed to reduce the stress level of the woman during the intraparty period. In the study, the pregnancy diagnosis form will be applied by the researcher to the pregnant women in the experimental and control group between the 28th and 36th weeks of the outpatient clinic. Visual Analog Scale will be applied to determine the Wijma Birth Expectation/Experience (W-DEQ A) Scale and birth fear in order to determine the birth fears of pregnant women in the 28th-36th week. During outpatient checks, the first saliva cortisol samples will be taken by the scholar Meserret Aslan between 8:30 and 09:00 in the morning. By Bursiyer Meserret Aslan, six hours of online pregnancy training will be given to the pregnant women in the experimental group and uninterrupted midwife support will be provided during the intrapartum period. After birth, mother and newborn saliva cortisol samples will be repeated by the scholar Meserret Aslan within the first half hour of the postpartum from the experimental and control groups. Before postpartum discharge procedures take place between 24th and 72nd hours, a sample of mother and newborn saliva cortisol will be taken and stored under appropriate conditions (Refrigerator (2-8 °C) 4 Days) by Meserret Aslan, a scholar from the experimental and control groups. The Birth Experience Scale and the wijma birth expectancy/birth experience (W-DEQ B) scale will also be applied before discharge. The world health organization's maximum acceptable cesarean section rate is 53.1%. Turkey has the highest cesarean section rate among OECD countries. There are studies that show that continuous midwife support in childbirth is useful in reducing the rate of cesarean sections. In addition, it is foreseen that reducing the stress levels of women and their babies who are offered uninterrupted midwife support will contribute to the prevention of mental illness in the postpartum period, which is one of the most fragile periods for women's mental health. Intrapartum continuous midwife support, which will facilitate adaptation to the role of mother in the postpartum period, will also contribute to the mother and baby bonding that form the basis of mental health in the future life of the baby. This study is expected to contribute to improving maternal and infant health, as well as improving public mental health. Evidence-based information will be provided to investigate saliva cortisol levels and to demonstrate the importance of intrapartum continuous midwife support in reducing stress levels of women and their babies.

ELIGIBILITY:
Inclusion Criteria:

* Women who can speak and understand Turkish.
* Women between the ages of 18 and 35.
* Women with their first pregnancy.
* Women with the only living fetus.
* Women who do not have any chronic diseases.
* Women who live with their spouses.
* Women who have not been diagnosed with risky pregnancy during pregnancy.
* Women whose pregnancy is between 28 and 36 weeks.
* Women who scored 38 or more on the Wijma Birth Experience/Expectation Scale A and agreed to participate voluntarily in the study.

Exclusion Criteria:

* Women who do not complete all the steps of the research.
* Those who develop any complications in the mother or baby during the birth process.
* Those who do not complete the research forms will be excluded from the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Saliva cortisol level | A salivary cortisol sample will be taken from each participant at the entrance to the delivery room. This evaluation will take 1 week.
  Saliva cortisol sample will be taken from prenatal pregnancy, mother and baby after birth to determine stress levels. The first saliva cortisol sample during pregnancy will be taken from the pregnant woman at the 28th-36th gestational week, and then the postpartum will be taken from both mother and baby within the first half hour. Finally, saliva cortisol test from mother and baby will be repeated within 24-72 hours before discharge.
Saliva cortisol level | A salivary cortisol sample will be taken from the mother and baby in the first half hour after birth. This evaluation will take 1 week.
  Saliva cortisol sample will be taken from prenatal pregnancy, mother and baby after birth to determine stress levels. The first saliva cortisol sample during pregnancy will be taken from the pregnant woman at the 28th-36th gestational week, and then the postpartum will be taken from both mother and baby within the first half hour. Finally, saliva cortisol test from mother and baby will be repeated within 24-72 hours before discharge.
Saliva cortisol level | A salivary cortisol sample will be taken from the mother and baby within 24-72 hours after birth. This evaluation will take 1 week.
  Saliva cortisol sample will be taken from prenatal pregnancy, mother and baby after birth to determine stress levels. The first saliva cortisol sample during pregnancy will be taken from the pregnant woman at the 28th-36th gestational week, and then the postpartum will be taken from both mother and baby within the first half hour. Finally, saliva cortisol test from mother and baby will be repeated within 24-72 hours before discharge.

SECONDARY OUTCOMES:
Level of fear of childbirth | The W-DEQ A scale will be applied to participants at least 12 weeks before birth. The W-DEQ B scale will be applied to participants within a maximum of 72 hours after birth. These evaluations will take 4 months.
  The W-DEQ-A scale will be applied in the prenatal period to determine the fear of childbirth. There are questions on the scale that include labor pains and how to feel, feelings when the baby is born, thoughts about childbirth within a month. It is planned to apply the W-DEQ-A scale to pregnant women who are in the 28th-36th week of pregnancy. In the postpartum period, the W-DEQ-B scale will be applied to determine the fear of childbirth. As the score increases, the fear of childbirth experienced by women increases. It is recommended to apply it at least 2 hours after birth and within 15 days at the latest. In this study, postpartum is planned to be applied within 24-72 hours.
Stress level | The Visual Analog Scale should have been administered to the participants at least 12 weeks before birth. This assessment will take 12 weeks.
  Visual Analog Scale (VAS) is a 10-point measurement tool and participants express the stress they perceive subjectively. This scale measures the stress that the person reports. "0" is expressed as not stressed at all, "10" is expressed as being stressed at the highest possible level.
Birth experience | The Birth Experience Scale will be applied to participants within a maximum of 72 hours after birth. This evaluation will take 12 weeks.
  The birth experience scale will be used to measure the birth experience. This scale is a 9-point self-assessment scale. The scale includes substances related to the birth experience and evaluates mothers' perception of stress, pain, control, fear and support during childbirth.It is planned to apply the birth experience scale to mothers within 24-72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Meserret ASLAN, Ankara, Altindağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/j.midw.2019.102535
- See also: Related Info — https://dx.doi.org/10.14744/zkmj.2021.73645
- See also: Related Info — https://doi.org/10.1016/j.neubiorev.2017.07.003
- See also: Related Info — https://doi.org/10.1186/s12884-019-2351-2
- See also: Related Info — https://doi.org/10.1097/aog.0000000000003748
- See also: Related Info — https://doi.org/10.1007/s00737-019-00968-2
- See also: Related Info — https://doi.org/10.1186/s12884-016-0798-y
- See also: Related Info — https://doi.org/10.1038/s41580-018-0068-0
- See also: Related Info — https://doi.org/10.1016/j.jpsychores.2017.09.002
- See also: Related Info — https://doi.org/10.1186/s12884-018-2069-6
- See also: Related Info — https://doi.org/10.1016/j.srhc.2019.06.004
- See also: Related Info — https://doi.org/10.1097/aog.0000000000001657
- See also: Related Info — https://doi.org/10.1017/s204017441800079x
- See also: Related Info — https://doi.org/10.1523/jneurosci.0733-19.2019
- See also: Related Info — https://doi.org/10.1186/s12913-020-05159-9
- See also: Related Info — http://dx.doi.org/10.1136/bmjopen-2019-030324
- See also: Related Info — https://data.oecd.org/healthcare/caesarean-sections.htm
- See also: Related Info — https://doi.org/10.1016/j.midw.2016.02.009
- See also: Related Info — https://doi.org/10.1016/s0140-6736(14)60789-3
- See also: Related Info — https://doi.org/10.1016/j.jogn.2015.12.008
- See also: Related Info — https://doi.org/10.1186/s12884-016-0944-6
- See also: Related Info — https://doi.org/10.1016/j.psyneuen.2018.09.031
- See also: Related Info — https://doi.org/10.1371/journal.pone.0230704
- See also: Related Info — https://doi.org/10.17179/excli2017-480